CLINICAL TRIAL: NCT03796793
Title: Developing Strategies for Effective Debridement in Patients for Venous Leg Ulcers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor & Chairman, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20180256; R01AR073614 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wound Edge Debridement Group (Experimental): Participants in this group will receive wound edge debridement in addition to standard of care (SOC) treatment for up to 4 weeks.
  Interventions: Procedure: Wound Edge Debridement; Other: Standard of Care Treatment
- Standard care group (Active Comparator): Participants in this group will receive only the standard care of treatment for up to 4 weeks.
  Interventions: Other: Standard of Care Treatment

INTERVENTIONS:
Procedure: Wound Edge Debridement — Wound debridement is performed using a sharp, circular disposable curette to remove the slough, non-viable tissue and any fibrous tissue down to the vascular base.
  Arms: Wound Edge Debridement Group
Other: Standard of Care Treatment — Standard of Care treatment will include foam dressing and 4 layer compression therapy, changed weekly.

SUMMARY:
The goal of this project is to use genomic profiling, candidate genes and proteins to develop guided surgical debridement to improve healing in chronic non-healing venous leg ulcers (VLUs) and to test the efficacy of this approach.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Conformation of venous disease by non-invasive venous studies with either Doppler-confirmed venous reflux, or having ≥ 2 clinical characteristics of venous insufficiency (varicose veins, lipodermatosclersosis, venous dermatitis, atrophie blanche, edema)
3. have a venous ulcer between the knee and ankle, at or above the malleolus
4. wound size would be greater than or equal to 5cm2 in area without exposed tendon, muscle or bone
5. wound duration of at least 6 months
6. VLU containing yellow/white slough with or without fibrous/scar tissue and/or non-viable tissue
7. ability of subject to tolerate limb compression bandage

Exclusion Criteria:

1. history of diabetes mellitus and a HbA1c > 12% (obtained within past 6 months)
2. Ankle brachial index(ABI) less than 0.80
3. any active cancer other than a nonmelanoma skin cancer; any previous cancer must be in remission for at least 5 years
4. suspicion of malignancy within VLU
5. life expectancy <6 months
6. history of kidney disease and creatinine greater than 2.0 (obtained within past 6 months)
7. history of liver disease and liver function test (ALT, AST, ALK PHOS, and bilirubin) >2x upper limit of normal (obtained within past 6 months)
8. requirement for long-term systemic corticosteroids or immunosuppressive therapy, or history of corticosteroid or immunosuppressive use in the 4 weeks prior to study entry
9. history of immunodeficiency
10. ulcers due to none venous etiology and leg ulcers associated with mixed etiology
11. Untreated osteomyelitis
12. Hepatitis
13. acute deep venous thrombosis
14. allergy to lidocaine and/or epinephrine
15. Subject's inability to successfully tolerate compression therapy that is changed weekly
16. Skin ulcer previously treated within the last 4 weeks with biologic therapies (e.g. cell therapy or growth factors)
17. if currently incarcerated
18. known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-03-18 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the genetic profile after debridement in the intervention group. | Baseline and 4 weeks
  RNA sequencing will be used to determine the number of differentially expressed genes of the intervention group in samples collected pre-debridement to samples collected post-debridement.

SECONDARY OUTCOMES:
Percent rate of healing | Up to 4 weeks
  Percent rate of healing is measured at every weekly visit and divided by 4 to calculate the average percent wound healing rate in cm2/week.

CONTACTS AND LOCATIONS:
Overall Officials: Marjana Tomic-Canic, PhD, Principal Investigator — University of Miami; Robert Kirsner, MD/PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No